CLINICAL TRIAL: NCT01296919
Title: New Insights on the Clinical Significance of the Uncinate Process Histopathology in Patients With Chronic Rhinosinusitis
Brief Title: The Clinical Significance of the Uncinate Process Histopathology in Chronic Rhinosinusitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Other Study IDs: AssutaHS10-2010037
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-02

CONDITIONS: Rhinosinusitis
Keywords: Chronic rhinosinusitis; Histopathology; Infundibulum; Lamina propria; Uncinate process
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathologic uncinate process tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sinus drainage: Adult patients with chronic rhinosinusitis who failed treatment with antibiotics and topical corticosteroids and underwent endoscopic sinus surgery. Preoperative evaluation included paranasal sinus CT scans. The diagnosis was confirmed by endoscopic examination showing purulent and/or mucopurulent discharge in the middle and/or superior meatus.

SUMMARY:
Given that the uncinate process is the gatekeeper of the sinuses, we hypothesize that inflammation of the uncinate process is associated with decreased ventilation and drainage of the paranasal sinuses and consequently with the inflammatory process occuring in the sinuses.

DETAILED DESCRIPTION:
The purpose of the present study is to gain insight into the histopathological changes of the uncinate process in patients with chronic rhinosinusitis through comparison of its mucosal and bony elements with those of the normal uncinate process without chronic inflammation (unpublished data: Gilead Berger, Ephraim Eviatar, Tatiana Kogan, Roee Landsberg).

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic rhinosinusitis who:

* Failed conservative medical treatment.
* Stopped treatment (topical or systemic corticosteroids) at least two months before endoscopic sinus surgery.
* Had a Lund-MacKay CT score of 2 and higher of 24 available.

Exclusion Criteria:

* Immunosuppressed patients.
* Patients in whom a pathologic evaluation of the middle turbinate was necessary (e.g., suspected neoplastic disorder).
* Patients with a Lund-MacKay CT score < 2 of 24 available.
* Pregnant women.
* Patients who underwent prior endoscopic sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis whose uncinate process had to be removed to enable surgical access to the sinuses.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Berger, MD, Principal Investigator — AssutaHS, Meir Medical Center; Eitan Yaniv, MD, Study Chair — Assuta Hospital Systems; Roee Landsberg, MD, Study Director — Assuta Hospital Systems
Locations (1):
- AssutaHS, Tel Aviv, Israel